CLINICAL TRIAL: NCT01128374
Title: The Effect of Non-Surgical Periodontal Therapy on Glycemic Control and Bacterial Levels in a Mexican-American Population With Type 2 DiabetesS
Brief Title: The Effect of Non-Surgical Periodontal Therapy on Glycemic Control and Bacterial Levels in a Mexican-American Population With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Isabel Gay, Assistant Professor - Periodontics, UT Houston Dental Branch, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UL1RR024148 (CTSA); UL1RR024148 (NIH)
Record Dates: First submitted 2010-05-20; First posted 2010-05-21 (Estimated); Last update posted 2013-01-15 (Estimated); Status verified 2013-01

CONDITIONS: Type 2 Diabetes Mellitus; Periodontal Disease
Keywords: Periodontal disease; Nonsurgical therapy; Type 2 Diabetes Mellitus; Bacterial burden; Gene polymorphisms
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Periodontal Diseases | interventions — Root Planing

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- intervention (Experimental): Therapy
  Interventions: Procedure: Periodontal Scaling and root planing

INTERVENTIONS:
Procedure: Periodontal Scaling and root planing — Participants will be instructed to brush their teeth using the modified Bass toothbrushing technique; the use of interproximal hygiene aids such as proximal brush or dental floss will be included. A full mouth scaling and root planning will be performed in 2 appointments (2 hours each) with the use of local anesthesia (typically 2% lidocaine with 1:100,000 epinephrine). In the control group, this treatment will be performed after all the data and samples have been collected and will encompass the last 2visits. Periodontal scaling and root planning treatment has been defined by The American Academy of Periodontology (AAP) as the standard of care for patients with periodontal disease. An ultrasonic instrument, scalers and curettes will be utilized to remove calculus and obtain a smooth root surface. The experimental subjects will be appointed 1 week later to complete the scaling and root planning procedure

SUMMARY:
Type 2 diabetes mellitus (T2DM) has become a significant pandemic with more than 7% of the population in the United States affected. Moreover, up to one-third of these individuals may not be aware of the diagnosis and, are not involved in treatment. In the Mexican-American population, prevalence rates may be up to 50%. Contributing factors such as poor education, low household income, language barriers and restricted access to medical services may increase this prevalence. The association between periodontal disease and diabetes has been well documented; however, interventional studies have resulted in conflicting conclusions on improvements in glycemic control following periodontal therapy.

Diabetes and periodontal disease share common pathways in pathogenesis, such as their polygenic nature and immunoregulatory dysfunction. To answer these questions, we, the investigators, propose this randomized controlled trial designed to elucidate how treatment of periodontal disease can be used for preventive and therapeutic purposes in a diabetic population as well as to study the role of IL-1 gene cluster polymorphisms as a risk factor for the presence of periodontitis in a Hispanic T2DM population. Our central hypothesis is that the Mexican-American T2DM population in Texas is at risk for an increased presence and severity of periodontal disease due to the presence of Il-1 gene cluster polymorphisms; furthermore we suggest that providing non-surgical periodontal therapy to this group will decrease the bacterial load associated with disease and as a consequence, will improve glycemic control as measured by HbA1c values. Our long-term goal is to study risk factors associated with the presence of periodontal disease and to understand how the treatment of periodontal disease can be used for preventive and therapeutic purposes in a Hispanic type 2 diabetic population.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years old
* Diagnosed type 2 diabetes mellitus
* Existence of moderate to severe periodontitis as defined by the American Academy of Periodontology
* In good general health - able to undergo the proposed therapy without compromise to existing health
* Demonstrated ability to read and understand written Spanish or English without the aid of ad-hoc interpretation by a third party
* Demonstrated ability to understand the proposed therapy and possible outcome
* Demonstrated willingness to comply with all protocol requirements as outlined in the informed consent document
* Willingness/ability to sign an informed consent document for their own inclusion in the study
* Hispanic origin as confirmed by patient records

Exclusion Criteria:

* Pregnancy at the time of enrollment (Pregnancy test is required for female study participants of child-bearing potential.)
* Use of antibiotics within last 3 months
* Immunocompromised health status
* Other medical conditions that represent a threat to life
* Osteoporosis
* Biphosphonates, corticosteroids or behavior alteration medications
* Historical abuse of alcohol or drugs
* Use of cigarettes/tobacco products within the past 12 months
* Mental diseases
* Any other oral pathology that compromise the patient's medical status
* Diagnosed type 1 diabetes mellitus (Information will be obtained from the medical records)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2010-06; Primary Completion 2012-09 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
HbA1c percentage | At baseline and 120 days after treatment

SECONDARY OUTCOMES:
microbial burden | Baseline and 120 days after therapy
gene polymorphisms | 120 days after enrolment

CONTACTS AND LOCATIONS:
Overall Officials: Isabel C Gay, DDS, MS, Principal Investigator — University of Texas Health Science Center Dental Branch; James Katancik, DDS, PhD, Study Chair — University of Texas Health Science Center at Houston Dental Branch; Gena Tribble, PhD, Study Director — University of Texas Health science Center Houston Dental Branch
Locations (1):
- The University of Texas Health Science Center Houston, Dental Branch, Houston, Texas, United States

REFERENCES:
- [Derived] Gay IC, Tran DT, Cavender AC, Weltman R, Chang J, Luckenbach E, Tribble GD. The effect of periodontal therapy on glycaemic control in a Hispanic population with type 2 diabetes: a randomized controlled trial. J Clin Periodontol. 2014 Jul;41(7):673-80. doi: 10.1111/jcpe.12268. Epub 2014 Jun 1. PMID 24797222